CLINICAL TRIAL: NCT03012867
Title: Effect of Different Enteral Nutrition Formulas on Glucose Homeostasis
Brief Title: Enteral Nutrition and Glucose Homeostasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marlene Wewalka, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUTR1
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Hyperglycemia Stress
Keywords: criticall illness; enteral nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fat-based (Active Comparator): Patients receive a fat-based enteral nutrition formula, which is routinely used as standard care in our ICU
  Interventions: Other: Diben, Fresenius Kabi
- glucose-based (Active Comparator): Patients receive a glucose-based enteral nutrition formula, which is routinely used as standard care in our ICU
  Interventions: Other: Fresubin original fibre, Fresenius Kabi

INTERVENTIONS:
Other: Diben, Fresenius Kabi — Patients receive Diben continously for 7 days
  Arms: fat-based
Other: Fresubin original fibre, Fresenius Kabi — Patients receive Fresubin original fibre continously for 7 days
  Arms: glucose-based

SUMMARY:
Different enteral nutrition formulas are tested on their effect on glucose homeostasis in critically ill medical patients.

DETAILED DESCRIPTION:
To assess whether enteral nutrition fomulas based either on fat or glucose influence glucose homeostasis differently in critically ill medical patients. All patients are admitted to a tertiary ICU and require mechanical ventilation.

Resting energy expenditure is assessed at baseline in the fasting state by indirect calorimetry. Total energy demand is calculated and patients are randomized to receive fat-based or glucose-based nutrition which is administered continously for 7 days. Indirect calorimetry is repeated on days 3 and 7 under continous nutrition. During the study period, various parameters of glucose homeostasis are assessed. Daily, there will be at least 3 measurements of blood glucose, more if the treating physician deems it necessary. Daily average glucose, daily glucose variability, overall area under the curve for glucose are calculated. Furthermore, energy intake by nutrition, medications (i.e. propofol), and glucose infusion, as well as substrate intake, and insulin demand per 24hrs are determined daily. Adverse effects such as episodes of hyper- or hypoglycemia, cholestasis, hypertriglyceridemia, diarrhea, vomiting, and the amount of gastric residual volume are noted.

ELIGIBILITY:
Inclusion Criteria:

* medical patient with need for mechanical ventilation
* FiO2 requirement < 60%
* need for nutritional support

Exclusion Criteria:

* contraindications against nutritional therapy
* hemodynamic shock (lactate of ≥ 4 mmol/l)
* severe hypertriglyceridemia (≥ 450 mg/dl)
* contraindications against enteral nutrion (intestinal obstruction, disruption or severe bleeding of upper gastrointestinal tract)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2014-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
average daily glucose | up to 7 days

SECONDARY OUTCOMES:
insulin demand per 24 hrs | up to 7 days
glucose variability | up to 7 days
nutrition-related side effects | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Zauner, MD, Principal Investigator — Medical University of Vienna, Department of Internal Medicine III, Division of Gastroenterology and Hepatology
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No